CLINICAL TRIAL: NCT07048548
Title: Assessment of Thyroid Hormone Levels and Potential Risk of Hypothyroidism in Healthcare Workers Exposed to Low-dose Ionizing Radiation
Brief Title: Assessment of THL and Potential Risk of Hypothyroidism in Healthcare Workers Exposed to Low-dose Ionizing Radiation
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/900
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid Function Monitoring
  Interventions: Behavioral: Thyroid Function Monitoring

INTERVENTIONS:
Behavioral: Thyroid Function Monitoring — This study will include healthcare professionals from the radiology and nuclear medicine departments at INMOL Cancer Hospital with at least one year of radiation exposure. A total of 44 participants will be selected through purposive sampling. Data will be collected using a structured questionnaire and blood tests for thyroid hormones (TSH, T3, T4) to assess thyroid function. Blood analysis will be conducted using CLIA or ELISA methods. The aim is to detect any association between low-dose radiation exposure and thyroid dysfunction.

SUMMARY:
"This study is designed to evaluate the thyroid health of healthcare workers exposed to low-dose ionizing radiation at INMOL Cancer Hospital, Lahore. Specifically, it investigates whether prolonged occupational exposure in radiology and nuclear medicine departments is associated with altered thyroid hormone levels or an increased risk of hypothyroidism. The thyroid gland is highly sensitive to radiation, and existing literature suggests a possible link between occupational exposure and thyroid dysfunction.

DETAILED DESCRIPTION:
A cross-sectional research design will be used over a four-month period. A sample of 44 participants will be selected using purposive sampling from the hospital's radiology and nuclear medicine staff.

ELIGIBILITY:
Inclusion Criteria:

* Staff members from radiology and nuclear medicine departments who meet both conditions.
* workplace experience exceeding one year
* age between 20 to 40 will be selected for this study.

Exclusion Criteria:

* Employees who have worked less than twelve months
* pregnant participants.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include healthcare professionals from the radiology and nuclear medicine departments at INMOL Cancer Hospital with at least one year of radiation exposure. A total of 44 participants will be selected through purposive sampling.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
thyroid function assessment | 12 Months
  Thyroid function is assessed through blood tests, primarily measuring TSH (Thyroid Stimulating Hormone), T4 (Thyroxine), and sometimes T3 (Triiodothyronine) levels. Abnormal levels of these hormones can indicate an underactive (hypothyroidism) or overactive (hyperthyroidism) thyroid.
  Normal Ranges (approximate):
  TSH: 0.4 - 4.0 mIU/L Free T4: 0.7 - 1.9 ng/dL Total T4: 5.0 - 12.0 μg/dL Total T3: 80 - 220 ng/dL

CONTACTS AND LOCATIONS:
Locations (1):
- INMOL hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No